CLINICAL TRIAL: NCT00398749
Title: Survey on the Treatment of Anemia Using Recombinant Human Erythropoietin 2
Brief Title: Survey on the Treatment of Anemia Using Recombinant Human Erythropoietin 2 (STAR-2)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR005596; EPOCAN4018
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; Neoplasms; Antineoplastic agents; Chemotherapy; Efficacy; Epoetin alfa
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Epoetin alfa: Epoetin alfa 40 000 IU once weekly variable treatment length
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — 40,000 IU once weekly, variable treatment length

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy (% response) of epoetin alfa in the treatment of anemia in adults receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
Anemia has been identified as a common complication and a widespread problem in the cancer population. Anemia is a condition in which a patient has below normal levels of hemoglobin, the substance in red blood cells that carries oxygen to all parts of the body. People with severe anemia may experience fatigue and shortness of breath with activity. Therefore, this condition can have a negative influence on a person's quality of life. Epoetin alfa, used to treat anemia in cancer patients, is a genetically engineered protein that stimulates red blood cell production. This study investigates treatment of anemia using epoetin alfa during chemotherapy in adult patients with cancer. The study is intended to collect information on normal medical practice and routine anemia management performed at the participating centers. This is an observational, non-randomized, prospective, comparative, parallel-group survey performed in The Netherlands. Patients with various severities of disease may enter the survey as soon as their epoetin alfa treatment starts and will be followed until the end of their epoetin alfa treatment. Patient data are collected in Case Report Forms (CRFs) until 4 weeks after the end of treatment with epoetin alfa. At the end of treatment completed CRFs will be collected. The assessment of effectiveness/response will be based on the following: cancer type and status, chemotherapy and other anti-cancer treatment, hemoglobin levels, use of blood transfusions, and serum iron levels and iron supplementation. Safety evaluations include the incidence of serious and non-serious adverse events. Because the study is observational, dosage, administration and duration of treatment is at discretion of treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of solid tumors, multiple myeloma (Kahlers' disease), non-Hodgkin lymphoma or Hodgkins' disease
* Patients must already be receiving chemotherapy or start their first cycle within a week of enrollment
* Patients must receive epoetin alfa treatment (expected treatment duration is at least 4 weeks)

Exclusion Criteria:

* Patients who cannot read the Dutch language and/or do not understand the Dutch Informed Consent Form and patients participating in either of our observational studies, EVALUATE or COMPARE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving epoetin alfa as anemia treatment during chemotherapy, as part of the common practice of participating physicians. Patients may enter the study as soon as their epoetin alfa treatment starts.
Sampling Method: Non-Probability Sample
Enrollment: 1927 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The assessment of effectiveness based on: epoetin alfa treatment schedule (dose and timing), hemoglobin effect, response to treatment (independent of blood transfusion), mean time to response, # of blood transfusions given, and iron supplementation | 4 weeks, 8 weeks and end of treatment

SECONDARY OUTCOMES:
Incidence of adverse events | from start epoetin treatment to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.

REFERENCES:
- See also: Survey on the Treatment of Anemia Using Recombinant Human Erythropoietin 2 (STAR-2) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=270&filename=CR005596_CSR.pdf